CLINICAL TRIAL: NCT02880202
Title: Impact of Massage Therapy on the Quality of Life of Hospice Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria I. Lapid, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-007515
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Pain; Anxiety; Depression; Quality of Life
Keywords: Massage Therapy; Hospice; Integrative Medicine; Palliative Care; Caregivers
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Massage Therapy (Other): Massage therapy for hospice patients.
  Interventions: Other: Massage Therapy

INTERVENTIONS:
Other: Massage Therapy — The massage therapy is provided by certified massage therapists and delivered in the home setting. Techniques and duration of massage therapy is customized based on input from the patient and/or caregiver at the start of the session regarding nature and location of discomfort and other symptoms, and based on other factors such as contra-indications/complicating factors, medical issues, and additional diagnoses. The number of massage therapy interventions range from 2-3, 1 week apart, with each session lasting between 20-45 minutes in duration.

SUMMARY:
This is a pilot study to evaluate the impact of massage therapy in hospice patients.

DETAILED DESCRIPTION:
As an integrative therapy, there is growing evidence that massage therapy can be an effective therapeutic tool for relief of pain and non-pain symptoms in hospice and palliative care patients. Massage therapy can provide comfort, relaxation, and improve quality of life for patients. The primary aim of the study is to gather data on the effects of complementary massage therapy on patient's symptoms and quality of life. The study goal is to improve patient symptoms of pain, anxiety, depression, and quality of life through the use of massage therapy provided to hospice patients. Questionnaires would be utilized before and after each massage intervention and would quantify symptom and quality of life levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Clinically determined by hospice staff to be appropriate for massage therapy (ESAS-r scores of 5 or greater on pain, depression, anxiety, or best well-being)
3. Place of residence within 30 minutes of downtown Rochester
4. Patient or caregiver must be able to participate in brief interviews and complete questionnaires (verbally or physically)

Exclusion Criteria:

1. Patients ineligible for massage therapy due to complexity of medical care including complex wound and multiple drains

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-08; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Edmonton Symptom Assessment System - Revised | Baseline to 3 weeks
  The primary endpoints are patient pain, depression, anxiety and wellbeing as measured by ESAS-r. Pro-rated area under the curve (AUC) statistics will be calculated for all individual items and total scores. The pro-rated AUC for ESAS-r measured pain, depression, anxiety, and wellbeing will all be utilized individually to assess the primary endpoint. The pro-rated AUC will be compared to the assessment score prior to any massage therapy. If there is any improvement, the massage therapy will be considered a success since any improvement will be seen as beneficial.

SECONDARY OUTCOMES:
Change in Edmonton Symptom Assessment System - Revised (Other symptoms) | Baseline to 3 weeks
  Secondary endpoints include all other symptoms (tiredness, drowsiness, nausea, lack of appetite, shortness of breath) as measured by the ESAS-r. Similar analysis will be conducted for all other endpoints as was conducted for the primary outcome. Pro-rated area under the curve (AUC) statistics will be calculated for all individual items and total scores.
Change in Linear Analogue Self Assessment (LASA) | Baseline to 3 weeks
  Secondary endpoints include symptoms as measured by the LASA (overall quality of life [QOL], mental well-being, physical well-being, emotional well-being, social activity, spiritual well-being, pain frequency, pain severity, fatigue, and social support). LASA items are stand alone, thus no scoring is necessary, but individual LASA items may be transposed so lower scores mean worse symptoms and higher scores mean less symptoms. This will allow consistency and thus easier data interpretation. Pro-rated area under the curve (AUC) statistics will be calculated for all individual items and total scores. Similar analysis will be conducted for all other endpoints as was conducted for the primary outcome.
Change in Patient Health Questionnaire for Depression and Anxiety (PHQ-4) | Baseline to 3 weeks
  Secondary endpoints include depression and anxiety symptoms as measured by the PHQ-4. Similar analysis will be conducted for all other endpoints as was conducted for the primary outcome.
Change in Pearlin role overload measure (ROM) | Baseline to 3 weeks
  Secondary endpoints include caregiver stress as measured by the ROM. Pro-rated area under the curve (AUC) statistics will be calculated for all individual items and total scores. Similar analysis will be conducted for all other endpoints as was conducted for the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Lapid, MD, Principal Investigator — Professor of Psychiatry
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No